Subject Identification

General Template Version Date: August 2016

Protocol Title: Dietary Restriction In Vascular Surgery

Principal Investigator: C. Keith Ozaki, MD

Site Principal Investigator:

Description of Subject Population: Adults undergoing selected vascular procedures involving an open major operation: carotid artery endarterectomy, aortic/iliac aneurysm repair, open lower extremity arterial procedures, major lower extremity amputation, or open hemodialysis access procedures

#### **About this consent form**

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

Partners HealthCare System is made up of Partners hospitals, health care providers, and researchers. In the rest of this consent form, we refer to the Partners system simply as "Partners."

If you have any questions about the research or about this form, please ask us. Taking part in this research study is up to you. If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

# Why is this research study being done?

This research study will compare the impact of dietary restriction pre-operatively compared to the standard nutrition that a patient typically eats before selected vascular surgery procedures major operation. We want to study how dietary restriction before surgery affects patient's response to surgery and recovery studies suggest that short-term dietary restriction may be beneficial before surgery. This study is a randomized, controlled mechanistic study physician at Brigham and Women's Hospital (BWH). This research has no external funding and is supported by the Division of Vascular and Endovascular Surgery at BWH.


Subject Identification


This study plans to enroll 80 research participants treated at BWH.

You are being asked to take part in this study because your doctor has recommended one of the following procedures:

- Carotid artery endarterectomy
- Aortic/iliac aneurysm repair (open, and endovascular if groin cut down planned)
- Open lower extremity arterial procedures (bypasses, aneurysm repair, arterial and bypass graft reconstructions)
- Major amputation of the lower extremity (below knee and above knee amputations)
- Open hemodialysis access procedures

Hydrogen sulfide has emerged as a critical gas signaling molecule in biological processes. Non-human scientific research published by the BWH vascular surgery research laboratory and others has linked hydrogen sulfide production to short-term dietary restriction. Dietary restriction means limiting what you eat (in this case excess protein and some calories) temporarily. Pilot data suggest that adverse post-operative outcomes like strokes, heart attacks, and wound healing problems may be modified by brief protein-calorie restriction in humans as well.

# How long will I take part in this research study?

If you choose to take part, you will be actively enrolled in the study for anywhere from 35 to 60 days.

# What will happen in this research study?

#### This is the visit/encounter schedule:

Visit 1: Baseline assessments (up to 30 days before your procedure)

Visit 2: Day of Surgery Visit 3: Post-operation day 1 Visit 4: Post-operation day 30

If you choose to take part in this study, we will ask you to sign this consent form before conducting any study procedures. We will review your medical history fully to ensure you qualify to safely participate in this research study. If you don't qualify, the study doctor will tell you why. After signing consent and you are determined to be eligible by a physician-investigator, you will be offered a taste test of the ScandiShake. This is a commercially available nutritional supplement used by people who need to gain weight. In this study it is being used to





achieve the dietary restriction diet. You will be able to choose which flavor you want if you are randomized to the restricted diet.

We will assign you by chance (like a coin toss) to the restricted diet group (called PCR), Group 1, or the control group, Group 2. The control group will be eating what they would normally and not changing their diet. You and the study doctor cannot choose your study group. You will have a 3 in 5 chance of being assigned to the restricted diet group. You will have a 2 in 5 chance of being assigned to the control group.

- Group 1: The restricted diet group will drink ScandiShake mixed with almond milk
- Group 2: Eats a normal, routine diet. You are encouraged to not change the way you eat.

Water intake is not restricted for either group, and participants should drink water as they normally do, and according to the pre-operative instructions given. Both diets can be consumed throughout the day and night.

If you do quality for the study, you will be asked to return to the Clinical Trials Hub (CTH) at BWH between 30 and 5 days before surgery for baseline assessments detailed below. This visit may be in conjunction with your anesthesia pre-operative evaluation, but may require an additional trip to the hospital. You will be asked to recall your diet the day before your baseline appointment and to record your diet for the four days before surgery and two weeks following the procedure. We will provide you with a free smartphone application called MealLogger, where you can document your food intake using pictures and directly talk to our licensed dieticians. If you do not have access to a smartphone, we can also provide a color-coded food diary to hand record meals.

The following are details related to each visit:

#### Visit 1: Baseline Assessments (Pre-operative Day 30-5)

- Collect information about your medical history, current health, and medications you are taking. We will also look at your medical record to help collect this information. To make sure this study is safe for you, you should be completely truthful with the study staff about your medical history.
- Physical exam, including height and weight.
- Blood Draw. This will be used for standard lab tests and measure production of stress and inflammation markers. We will draw about 35mL of blood (about 2.5 tablespoons).
- If you are female who is of children bearing potential, blood will be drawn and tested to ensure you are not pregnant. If you are pregnant, you cannot take part in this study.





- Download and review the MealLogger phone application, where you will be able to document your diet with pictures that are automatically shared with our licensed dietician who can respond with clarifications about what you have eaten. You will be asked to record what your dietary intake four days before admission, and every day after surgery until post-operative day 14.
  - If you cannot use the MealLogger app, we will give you a color-coded food diary to hand record meals.
- We will ask for a 24-hour food recall, to gather a baseline assessment of your typical diet.
- Randomization to a diet group. If randomized to the dietary restriction group, we will supply you with the ScandiShakes at this visit to eat for the 4 days leading up to your surgery. We will allow you to sample the flavors, so you can choose your preference.

#### **Visit2: Day of Surgery**

The day of surgery will ask you to provide a repeat blood draw for research purposes, which will be done at the same time as blood draws needed for your care. During the surgery, a small tissue sample will be collected by your surgeon for analysis, about the size of an eraser head. From this point on, you may resume your usual diet according to standard post-operative care, regardless of what diet you were assigned to. We will still ask you to continue logging your diet using either MealLogger or paper record.

At this visit, we will collect/perform:

- Blood sample
- Weight
- Food diary (if applicable)
- Fat tissue samples will be taken and analyzed. These samples will each be about the size of the eraser head of a pencil.
- Discarded tissue that might be left over after your surgery will also be collected for analysis.

#### **Visit 3: Post-Operation Day 1**

Based on your recovery progress, your surgery team will determine when you will be discharged from the hospital. We will see you in the hospital on post-operation day 1 for the following procedures. Both groups (PCR diet and normal diet) will resume normal diet immediately after surgery according to recommendation by the clinical team. For subjects who do not need an overnight hospital stay, this visit will occur after surgery but before you are discharged.


| Subject Identification |
|------------------------|


At this visit, we will collect/perform:

- Physical exam
- Blood Sample
- Collect the appropriate food diary entries if not using MealLogger app

#### Visit 4: 1-Month Post-Operative Research Study Visit (Day 30 +/- 2 weeks)

You will return to the hospital for a standard post-operative evaluation with your vascular surgeon. At the end of this visit, your study participation will end.

At this visit, we will collect/perform:

- Physical exam
- Wound evaluation of the incision
- Information about any changes in your health, procedures since your surgery, or problems you have had
- Collect the appropriate food diary entries if not using MealLogger app (for two weeks post-op)
- End of study survey about your opinions and experience with the trial

At the one-year mark after your surgery, we will review your medical record at to record any clinically important events.

#### **Unscheduled Visits**

If you have any side effects from your surgical care, your doctor may request that you come in for an unscheduled visit for further assessment of the side effect.

#### **Future Use of Stored Specimens**

The small amount of blood at Visits 1-3 will be labeled with a code number (not your name) and temporarily stored and analyzed for chemical composition in a vascular research laboratory at BWH. Samples will also be stored and analyzed in The Mitchell Laboratory (Harvard School of Public Health) and by Dr. Karen Ho (Northwestern Feinberg School of Medicine). Fat samples will be studied at BWH for chemical composition and microscopic examination. These will be analyzed at BWH for the effects of diet on lipid composition, and inflammatory markers predictive of the response to surgical stress. The key to the code connects your name to your samples and health information. The study doctor and coordinators will keep the key to the code in a password locked file on a Partners secured computer.

Additionally, discarded tissue specimens will be examined microscopically at BWH. Enrolled patients and their clinical data will be entered into a study-specific database.


# Partners HealthCare System Research Consent Form General Template Version Date: August 2016 Subject Identification

Do you agree to let us store discarded tissues and adipose samples for histology study (under the microscope)?

| ( ) YES ( ) NO Initials |
|-------------------------|
|-------------------------|

# What are the risks and possible discomforts from being in this research study?

Your doctor will explain the risks of the medical procedure (carotid endarterectomy, aortic/iliac aneurysm repair, lower extremity arterial revascularization, major lower extremity amputation or open hemodialysis access procedures) you are having. Your doctor will ask you to sign a separate clinical consent form that explains the risks and benefits of the procedure. Allowing your leftover samples to be used for research will not change the risks of the medical procedure.

At this time, there are no known medical risks associated to short-term PCR diets. We have successfully completed a pilot study here at BWH investigating and confirming the safety of the PCR diet before vascular surgery.

However, as a result of taking part in this study, you are at risk for the following side effects. You should discuss these with the study doctor and your regular health care provider.

### **Risks of Blood Drawing**

You may have a bruise (a black and blue mark) or pain where we take the blood samples. There is also a small risk of infection, lightheadedness, and/or fainting.

#### Risks of Pregnancy and Information about Birth Control

The effect of dietary restriction on an embryo or fetus (developing baby still in the womb), or on a breastfeeding infant, is unknown and may be harmful. Because of these unknown risks, women cannot take part in this study if they are:

- Pregnant
- Trying to become pregnant
- Breastfeeding

If you are a menopausal woman and have not had a period for the past 12 months or more, you will not need to have a pregnancy test. Also, if you have had any well-documented method of surgical sterilization, you will not need to have a pregnancy test. Methods of surgical sterilization


Subject Identification


include having had a hysterectomy (removal of the uterus with or without the ovaries), bilateral oophorectomy (removal of both ovaries), a tubal ligation (having your tubes tied), or transvaginal occlusion (plugging the opening of the tubes with a coil). All other female subjects must have a negative pregnancy test.

If you are a female who is able to become pregnant and you decide to take part in this study, you must have a negative pregnancy test at the screening visit (Visit 1), and you must agree to use birth control for at least 4 weeks after surgery.

Acceptable birth control methods for use in this study are:

- Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
- Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- Intrauterine device (IUD)
- Abstinence (no sex)

#### Fat (Adipose) Biopsies

Adipose (fatty tissue) biopsies (sample of tissue taken from the body to examine it more closely) add about 30-60 seconds more to your surgery but hold no other known risks.

#### Infection

Infection is a risk of any surgery, including the one you are having.

#### **New Findings**

Sometimes during the course of a research study, we get new information that affects the risks of taking part in the study. We will tell you about any new information that might change your decision to be part of this study or continue taking part. You may contact the study doctor or any member of the study team at any time after you complete taking part in the study to find out if any new information about this study has become available.

#### **Inconveniences to You**

Taking part in a research study can be inconvenient. Please think about the time commitments and responsibilities you will be agreeing to as a research subject. You must carefully follow any instructions given to you.

Additional visit to the hospital: We ask that you come to the hospital for one visit that may not be standard of care, Visit 1 (between 30-5 days before surgery). Any time spent in the hospital can be stressful.





#### **Possible Hunger**

If you are assigned to the restricted diet you may experience hunger or discomfort. If you feel too hungry or uncomfortable you may choose to resume a normal diet while recording all intake and stay in the study. You may also withdraw at any time.

#### **Possible Fatigue**

You may also experience fatigue pre-operatively if randomized to the restricted diet.

## What are the possible benefits from being in this research study?

You may or may not benefit medically from taking part in this study. We hope that if you receive the restricted diet you may have less chance of complications after your surgery, but this is unproven. We do not expect any benefit if you are randomized to the non-dietary restricted arm.

Choosing to take part in this research study may help others having surgery in the future. It is important to know that you may <u>not</u> receive any direct benefit from participating.

## What other treatments or procedures are available for my condition?

You do not have to take part in this study to be treated for your medical condition. You can have the procedure done without electing to be a part of this study. You should discuss these choices with your doctor.

# Can I still get medical care within BWH if I don't take part in this research study, or if I stop taking part?

Yes. Your decision won't change the medical care you get within BWH now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

# Can I still get medical care within Partners if I don't take part in this research study, or if I stop taking part?

Yes. Your decision won't change the medical care you get within Partners now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.





Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. We will tell you if we learn new information that could make you change your mind about taking part in this research study.

# What should I do if I want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

# Will I be paid to take part in this research study?

Yes, you will be paid \$50 for completing the baseline study visit, \$50 for successfully recording your 4-day dietary intake before surgery, and \$100 for successfully completing the end of study visit for a total of \$200. We will also provide a parking voucher for the baseline visit.

We will not pay you for missed or incomplete visits. We will pay you by check, so please allow time for processing. We will ask you to provide your social security number for reimbursement purposes.

You will also receive a complimentary custom cooler bag.

# What will I have to pay for if I take part in this research study?

The Division of Vascular and Endovascular Surgery at Brigham and Women's is providing the PCR diet and all research tests at no additional cost to you.

Although study funds will pay for certain study-related items and services, we will bill your health insurer for your surgery, anesthesia, and the routine items and services you would have received even if you did not take part in the research.

Your surgery and the overnight post-operation stays are not part of this study. The costs related to your surgery and for any routine care related to that surgery will be billed to you or your insurance company in the usual way.


Subject Identification


You will be responsible for payment of any deductibles and co-payments required by your insurer for this routine care or other billed care. If you have any questions about costs to you that may result from taking part in the research, please speak with the study doctors and study staff. If necessary, we will arrange for you to speak with someone in Patient Financial Services about these costs.

# What happens if I am injured as a result of taking part in this research study?

We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the next section of this consent form.

# If I have questions or concerns about this research study, whom can I call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

Dr. C. Keith Ozaki is the person in charge of this research study at BWH. You can call him at (857)-307-1920, Monday-Friday 8:30am – 5:00pm. You can also call any Vascular Surgery Clinical Research Assistant at (617) 525-8555, Monday-Friday 8:00 a.m. – 5:00 p.m. with questions about this research study or any research related concerns you may have.

If you have questions about the scheduling of appointments or study visits at BWH, call the Vascular Surgery Research Team at (617)-525-8555 or the Vascular Surgery Administrative team at (857)-307-1920.


Subject Identification

**General Template** 

**Version Date: December 2008** 

If you want to speak with someone **not** directly involved in this research study, please contact the Partners Human Research Committee office. You can call them at 857-282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research

Also, if you feel pressured to take part in this research study, or to continue with it, they want to know and can help.

# If I take part in this research study, how will you protect my privacy?

During this research, identifiable information about your health will be collected. In the rest of this section, we refer to this information simply as "health information." In general, under federal law, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use, and share your health information for research and why they may need to do so.

#### In this study, we may collect health information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires

# Who may see, use, and share your identifiable health information and why they may need to do so:

- Partners research staff involved in this study
- The sponsor(s) of this study, and the people or groups it hires to help perform this research
- Other researchers and medical centers that are part of this study and their ethics boards
- A group that oversees the data (study information) and safety of this research
- Non-research staff within Partners who need this information to do their jobs (such as for treatment, payment (billing), or health care operations)
- The Partners ethics board that oversees the research and the Partners research quality improvement programs.
- People from organizations that provide independent accreditation and oversight of hospitals and research


| Subject Identification |
|------------------------|


- People or groups that we hire to do work for us, such as data storage companies, insurers, and lawyers
- Federal and state agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health, and other US or foreign government bodies that oversee or review research)
- Public health and safety authorities (for example, if we learn information that could mean harm to you or others, we may need to report this, as required by law)
- Other:

Some people or groups who get your health information might not have to follow the same privacy rules that we follow and might use or share your health information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your health information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your health information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your information for any mailing or marketing list. However, once your information is shared outside Partners, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your health information.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifying information **will not** be used for these purposes without your specific permission.

# **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your health information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your health information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others.


| Partners HealthCare System<br>Research Consent Form | | |
|---|---|---|
| General Template Version Date: August 2016 | | Subject Identification |
| You have the right to see and get a copy of your treatment or for payment. To ask for this inform research study. You may only get such informat | ation, please con | tact the person in charge of this |
| <b>Informed Consent and Authorizat</b> | ion | |
| Statement of Person Giving Informed Consen | t and Authoriza | tion |
| <ul> <li>I have read this consent form.</li> <li>This research study has been explained to any), other possible treatments or proceded.</li> <li>I have had the opportunity to ask question.</li> <li>I understand the information given to me.</li> </ul> | ures, and other in | |
| Signature of Subject: | | |
| I give my consent to take part in this research stube used and shared as described above. | dy and agree to a | allow my health information to |
| Subject | Date | Time (optional) |
| Signature of Study Doctor or Person O | S | ent: |
| Statement of Study Doctor or Person Obtaining | ng Consent | |
| <ul> <li>I have explained the research to the study</li> <li>I have answered all questions about this r</li> </ul> | = | the best of my ability. |
| Study Doctor or Person Obtaining Consent | Date | Time (optional) |


IRB Protocol No: 2018P002133 Consent Form Valid Date: 6/10/2019

**Sponsor Protocol No: NA** IRB Amendment No: AME7

Sponsor Amendment No: N/A

IRB Amendment Approval Date: 6/7/2019

Consent Form Expiration Date: 11/21/2019

| Partners HealthCare System<br>Research Consent Form | | |
|---|---|---|
| General Template | | Subject Identification |
| Version Date: August 2016 Consent of Non-English Speaking S | Subjects Using the | "Short Form" in the |
| Subject's Spoken Language | | |
| Statement of Hospital Medical Interpret<br>As someone who understands both English<br>in the subject's language, the researcher's properties are given the opportunity to ask questions. | and the language spok<br>resentation of the Engl | |
| Hospital Medical Interpreter | Date | Time (optional) |
| OR Statement of Other Individual (Non-Inter As someone who understands both English that the English version of the consent form own language, and that the subject was given | and the language spok<br>was presented orally | to the subject in the subject's |
| Name | | Time (optional) |

Consent Form Version: 06/06/2019


Consent Form Title: DRIVeS ICF Update\_CLEAN\_06JUN2019 IRB Protocol No: 2018P002133 Consent Form Valid Date: 6/10/2019 Consent Form Expiration Date: 11/21/2019

Sponsor Protocol No: NA IRB Amendment No: AME7

Sponsor Amendment No: N/A